CLINICAL TRIAL: NCT00204555
Title: A Randomized Open Label Study to Evaluate the Safety and Efficacy if Imiquimod 5% Cream Applied 3 Times Per Week for 8 or 12 Weeks in the Treatment of Low Risk Nodular Basal Cell Carcinoma
Brief Title: Safety and Efficacy Study of Imiquimod 5% Cream Applied 3x Per Week for 8 or 12 Weeks in Low Risk Nodular Basal Cell Carcinoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BCC-IMI-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2007-04

CONDITIONS: Carcinoma, Basal Cell
Keywords: nodular basal cell carcinoma; Imiquimod; topical treatment; Adjuvants, Immunologic; Antineoplastic Agents; Interferon Inducers
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

INTERVENTIONS:
Drug: Imiquimod

SUMMARY:
Results from a pilot study demonstrated that topical imiquimod could clear superficial and nodular BCCs. Three phase II dose response studies in subjects with nodular BCC (nBCC) showed that the histological cure rates with imiquimod depend on the doses applied per week and the duration of treatment. Daily dosing or 5 times per week applications showed higher total clearance rates than 3 times per week dosing or less frequent dosing. Furthermore, a 12 week treatment period resulted in better efficacy results than a duration of only 6 weeks. On the other hand, local skin reactions increased with the doses applied per week. So a prolonged treatment period of 8 or 12 weeks with an application frequence of 3 times a week seems to be a good compromise between efficacy and safety.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is a malignant skin cancer that is believed to develop from the basal layer of the epidermis. Ultraviolet (UV) radiation is the primary cause of BCC. It induces local and systemic immuno-suppression, p53 mutations, pyrimidine covalent dimers in desoxyribonucleic acid (DNA), and bcl-2 overexpression. All of these UV-induced changes are believed to be critical in the pathogenesis of BCC.

Topical application of imiquimod induces local interferon-alpha (IFN-alpha), interleukin-12 (IL-12), and tumor necrosis factor-alpha (TNF-alpha), with a resulting cytokine cascade that may induce and/or support a cytotoxic T-lymphocyte (Th1) immune response. Intralesional IFN-alpha has been shown to be effective for the treatment of BCC. Imiquimod may be an effective therapy for BCC.

Results from a pilot study demonstrated that topical imiquimod could clear superficial and nodular BCCs. Three phase II dose response studies in subjects with nodular BCC (nBCC) showed that the histological cure rates with imiquimod depend on the doses applied per week and the duration of treatment. Daily dosing or 5 times per week applications showed higher total clearance rates than 3 times per week dosing or less frequent dosing. Furthermore, a 12 week treatment period resulted in better efficacy results than a duration of only 6 weeks. On the other hand, local skin reactions increased with the doses applied per week. So a prolonged treatment period of 8 or 12 weeks with an application frequence of 3 times a week seems to be a good compromise between efficacy and safety.

The current safety and efficacy study of imiquimod 5% cream in the treatment of nodular basal cell carcinoma (nBCC) will use a composite endpoint including both a clinical (visual) assessment of the target tumor site and a histological evaluation of an excisional surgery taken from the target tumor site for primary assessment of complete tumor clearance 8 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to understand and willing to give informed consent prior to study procedures
* Age 18+
* Have one BCC which meets the following criteria: a primary tumor (not recurrent, not previously biopsied or treated; non-infected; located on the limbs, trunk (anogenital area excluded), neck, or head. The target tumor must be visible; maximum tumor area of 1.5 cm in diameter; macroscopically (clinically) consistent with nodular BCC; nodular subtype, with circumscribed growth pattern; histologically consistent with nBCC, and having no histological evidence of aggressive growth patterns; easily identifiable and treatable by subject or reliable subject representative;
* Are willing and able to participate in the study as an outpatient, making necessary visits to the clinic during the treatment period and comply with study requirements, including the following: A minimum of 1 and a maximum of 3 prestudy confirmatory biopsies of different tumors before beginning study drug treatment (each biopsy will remove no more than 25% of the target tumor); at least 4 or 5 clinic visits during the study; blood sampling at screening/initiation visit and end of treatment; urine pregnancy testing for females of childbearing potential at the screening/initiation visit and the end of treatment visits
* Are free of any significant physical abnormalities at the potential application site area, which would interfere with assessment of possible site reactions (eg, eczema, psoriasis, tattoos)
* If female and of childbearing potential, has negative urine pregnancy tests during screening/initiation visit, and is willing to use a medically acceptable method of contraception during the treatment period

Exclusion Criteria:

* High-risk areas within 0.5 cm of the eyes
* Have evidence of clinically significant, unstable medical conditions such as metastatic tumor or tumor with high probability of metastatic spread, cardiovascular (NYHA class III, IV), immunomodulation or immunosuppressive therapies, hematologic, hepatic, renal, neurologic, endocrine, collagen-vascular, gastrointestinal
* Have or had other malignant tumors of the skin within the target tumor site or surrounding area (eg, malignant melanoma, epithelioma spinocellular, squamous cell carcinoma). The surrounding area includes the skin within 2 cm of the target site margins in all directions
* Have received the following treatments for any indication in the target tumor site or surrounding area within the designated time period (6 weeks) before treatment initiation: Topical retinoids, Topical steroids, Surgical excision, Curettage, Cryo-, Thermo- or Chemodestruction, Photodynamic therapy, Therapeutic UV-Radiation
* Have received the following systemic treatments within the designated period before study treatment initiation: Interferon (6 weeks), Immunomodulators or immunosuppressive therapies (10 weeks), Cytotoxic drugs (6 months), Investigational drugs (8 weeks), Drugs known to have major organ toxicity (8 weeks), Corticosteroids (oral or injectable) (6 weeks), Inhaled corticosteroids (>1200 ng/day for beclomethasone, or >600 ng/day for fluticasone)(4 weeks)
* Have received any systemic cancer chemotherapy within 6 months before study treatment initiation
* Have known allergies to any excipient in the study cream (isostearic acid, benzyl alcohol, cetyl alcohol, stearyl alcohol, polysorbate 60, sorbitan monostearate, white petrolatum, glycerin, methyl paraben, propyl paraben, purified water, and xanthan gum
* Are known to be pregnant or lactating (currently or within the past 3 months). If the subject was pregnant, at least 3 months must have elapsed since parturition or termination
* Have any dermatological disease in the target tumor site or surrounding area that may be exacerbated by treatment with imiquimod or cause difficulty with examination (eg psoriasis, eczema)
* Are currently or within the past 8 weeks participating in another clinical study
* Have active chemical dependency or alcoholism as assessed by the investigator
* Have had a systemic bacterial or viral infection within 2 weeks prior to study initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-01; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the clearance rate, defined as the proportion of subjects who are clinically and histologically clear of BCC at the treated nodular BCC target tumor site at the 8 week post-treatment visit

SECONDARY OUTCOMES:
intensity of local skin reactions such as erythema, vesicles, scarring | every 4 weeks during treatment
Cosmetic outcome | 8 weeks posttreamnt

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, MD, Principal Investigator — Skin Cancer Program, Department of Dermatology, University Hospital Tübingen
Locations (1):
- Skin Cancer Program, Department of Dermatology, Liebermeisterstrasse 8, Tübingen, Baden-Wurttemberg, Germany